CLINICAL TRIAL: NCT05976971
Title: Microstructural Brain MRI Biomarkers in Patients With Idiopathic REM Sleep Behaviour Disorder at 7 Tesla
Brief Title: Microstructural and Sodium 7 Tesla Brain MRI in Idiopathic REM Sleep Behaviour Disorder
Acronym: SODISLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Aix Marseille Université (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM22_0397; ID-RCB (Other: 2023-A00457-38)
Record Dates: First submitted 2023-07-12; First posted 2023-08-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: REM Sleep Behaviour Disorder
Keywords: 7T MRI; Parkinson's disease; synucleinopathies
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease; Synucleinopathies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with REM Sleep Behaviour Disorder (Other)
  Interventions: Other: 7T MRI
- Healthy volunteers (Other)
  Interventions: Other: 7T MRI

INTERVENTIONS:
Other: 7T MRI — Subjects will have a 7T MRI and questionnaires on the only day of clinical study.
  Other Names: Questionnaires

SUMMARY:
By 2030 the number of patients with Parkinson's Disease (PD) would increase by 56% affecting 1 out of 120 people older than 45 years-old. It is known that 10-15 years before the onset motor symptoms such as tremor, rigidity and akinesia, patients often experience a specific sleep trouble called REM sleep behaviour disorder (RBD). Follow-up of those subjects showed there was a conversion rate to PD and related disorders (called synucleinopathies) over 80%.

The pathophysiology of RBD is poorly understood. The development of cutting-edge technologies such as 7 Tesla MRI and the optimisation of image processing methods made it possible to non-invasively explore in vivo small brain structures involved in sleep and movement disorders.

The investigators hypothesize that brain and brainstem microstructure, composition, sodium homeostasis and connectivity may change in 15 isolated RBD (iRBD) subjects compared with 15 healthy controls and that these changes may be correlated with clinical scores.

This study would help fill the gap in early diagnosis of synucleinopathies, by contributing to better targeting patients who could be included in therapeutic trials with a neuroprotective effect. Besides, the exploration of original pathophysiological pathways such as sodium homeostatis could provide the necessary arguments for the development of new target therapeutics.

ELIGIBILITY:
Inclusion Criteria for patients with REM Sleep Behaviour Disorder :

* Patient aged between 40 and 80 years old
* Patient fulfilling the diagnostic criteria for RBD (International Classification of Sleep Disorders version 3, American Academy of Sleep Medicine, 2014) with polysomnographic confirmation (which will be carried out as part of the routine work-up);
* UPDRS Part III score under or equal to 5
* The patient is enrolled in the French social security system
* The patient understood and signed the consent to participate in the study.

Inclusion Criteria for control group :

* Patient aged between 40 and 80 years old
* Score under or equal 4 for the RBD screening questionnaire
* UPDRS Part III score under or equal 5
* The patient is enrolled in the French social security system
* The patient understood and signed the consent to participate in the study.

Exclusion Criteria :

* Patient / Subject with a history of central nervous system disease (e.g. PD, Alzheimer's disease, stroke, brain tumour, multiple sclerosis, amyotrophic lateral sclerosis, etc.). If a doubt exist, this criterion will be left to the judgement of the principal investigator, who is a neurologist.
* Contraindications to 7T MRI: presence of a metal in the body or in the eye, patient with a pacemaker or neurostimulator, cochlear implants or any implanted electronic medical equipment in general, metallic heart valve, aneurysm clips.
* Claustrophobia.
* Montreal Cognitive Assessment Test (MOCA) < 25/30
* Pregnant or breast-feeding woman or protected person (under guardianship, curatorship, deprived of liberty).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
3D cartography the rate of difference of atrophy between the idiopathic REM Sleep Behaviour Disorder (iRBD) and control subjects | Time of the Inclusion
  Voxel based morphometry evaluated with Matlab and SnPM
3D cartography difference of neuromelanin between the iRBD and control subjects with T1 sequence | Time of the Inclusion
  Neuromelanin contrast ratio
3D cartography difference of neuromelanin between the iRBD and control subjects with Magnetization transfert sequence | Time of the Inclusion
  Magnetization transfert contrast ratio
3D cartography the rate of difference of Quantitative Susceptibility Mapping between the iRBD and control subjects | Time of the Inclusion
  Iron load evaluation in ppb
3D cartography difference of Mean diffusivity between the iRBD and control subjects | Time of the Inclusion
  Mean diffusivity in mm2/s
3D cartography difference of Fractional anisotropy between the iRBD and control subjects | Time of the Inclusion
  Fractional anisotropy between 0 and 1

SECONDARY OUTCOMES:
3D cartography difference of total sodium concentration between the iRBD and control subjects | Time of the Inclusion
  total sodium concentration in mmol/L acquired with a specificic MRI coil
3D cartography difference of structural brain connectivity between the iRBD and control subjects | Time of the Inclusion
  A network-based statistics analysis will be performed: from Diffusion tensor imaging, a connectivity matrix will be populated for each subject. A t-test contrasting the two groups (iRBD and control subjects) will then be computed for each pairwise association. Finally, permutation testing will be used to ascribe a p-value controlled for the family-wise error rate to each connected component based on its size.
Rate of Dependency between MRI parameters and demographic data | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the age and MRI parameters
Rate of Dependency between MRI parameters and demographic data | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the sex and MRI parameters
Rate of Dependency between MRI parameters and demographic data | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the laterality and MRI parameters
Rate of Dependency between MRI parameters and demographic data, clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the MDS-UPDRS I (Movement disorders society - Unified Parkinson's Disease Rating Scale) scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the MDS-UPDRS II scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the MDS-UPDRS III scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the SCOPA-AUT scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the HAD scale (Hospital Anxiety and Depression scale) and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the RBD (Rem sleep behaviour disorder) and MRI parameters
Rate of Dependency between MRI parameters and demographic data, clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the Pittsburgh sleep quality index and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the Starkstein motivation scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the non motor fluctuation scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the MoCA scale and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the phonemic and category fluencies and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the Benton judgement of lines and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the quality of life SF-36 and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the Miami Hallucinations questionnaire and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the treatement intake and MRI parameters
Rate of Dependency between MRI parameters and clinical scores/questionnaires | Time of the Inclusion
  Pearson, Spearman or logistic regression, depending on the blood pressure test and MRI parameters

CONTACTS AND LOCATIONS:
Overall Officials: Francois Cremieux, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance - Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No